CLINICAL TRIAL: NCT07235397
Title: Evaluating the Benefits Of RSV MaternaL vAccination Using a Scottish National Dataset.
Acronym: BORLAND
Status: Not yet recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C3671083
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-10

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — abrysvo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Exposed: Infants whose mother received ABRYSVO vaccine during pregnancy 14 days or more before delivery
  Interventions: Biological: ABRYSVO
- Unexposed: Infants born to mothers who did not receive ABRYSVO during pregnancy will be considered unexposed

INTERVENTIONS:
Biological: ABRYSVO — ABRYSVO
  Groups: Exposed

SUMMARY:
This study will use a retrospective cohort design and will be conducted within routinely collected national healthcare and statutory demographic datasets held by PHS and National Records of Scotland (NRS). As such, there will be no active enrollment of study participants, no direct contact with study participants, no collection of any primary data outside of the standard of care (SOC), and no requirement for informed consent.

This study design was chosen due to several advantages, over other possible designs, including the ability to evaluate incidence of study outcomes in exposed and unexposed infants, ability to follow infants longitudinally to evaluate study outcomes through 12 months of age, and ability to evaluate all-cause outcomes.

Study endpoints, including RSV-associated LRTD hospitalization and RSV-associated hospitalization, among infants born to ABRYSVO-vaccinated mothers (exposed group) will be compared with those among infants born to ABRYSVO-unvaccinated mothers (comparison group) initially from birth through 6 months of age, with later analysis from birth through 12 months as the infants reach this age threshold and their data become available.

ELIGIBILITY:
Infants must meet all inclusion criteria to be eligible for inclusion in the study:

1. Live birth in Scotland from 1st September 2024 to 28th February 2026
2. Gestational age at birth ≥28(0/7) weeks of gestation (earliest gestational age eligible for ABRYSVO vaccination)

Infants meeting any of the following criteria will not be included in the study:

1. Born to a mother who received any licensed or investigational RSV vaccine other than ABRYSVO at any time during pregnancy
2. Meets UK national guidelines for monoclonal antibody receipt

Ages: 0 Years to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This will be a whole population birth cohort study of all live-born infants born in Scotland during the study period. In Scotland, all infants are assigned a unique identifier, the Community Health Index (CHI) at birth. CHI is a common identifier across all National Health Service (NHS) healthcare encounters and allows linkage of all healthcare data to statutory datasets such as death records. The patient population will include all live-born infants born in Scotland over an 18-month accrual period, from 1st September 2024 - 28th February 2026 (or end of RSV season) and their mothers (approximately 69,000 mother-infant pairs). Selection criteria for the population were based on the time period of the RSV season in Scotland and the earliest gestational age eligible for ABRYSVO vaccination, per the MHRA. All infants will be followed for 12 months after birth; thus, the last outcome assessment will be approximately 28th February 2027.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
PCR-confirmed RSV-associated LRTD hospitalization occurring ≤180 days after birth (first episode) | ≤180 days after birth

SECONDARY OUTCOMES:
PCR-confirmed RSV-associated hospitalization occurring ≤180 days after birth (first episode) | ≤180 days after birth
PCR-confirmed RSV-associated LRTD hospitalization occurring ≤180 days after birth (first episode) stratified by term/preterm status and by gestational age at vaccination | ≤180 days after birth
PCR-confirmed RSV-associated hospitalization occurring ≤180 days after birth (first episode) stratified by term/preterm status at delivery and by gestational age at vaccination | ≤180 days after birth
PCR-confirmed RSV-associated LRTD hospitalization occurring ≤360 days after birth (first episode) (by cumulative and by discrete age-intervals) | ≤360 days after birth
PCR-confirmed RSV-associated hospitalization occurring ≤360 days after birth (first episode) (by cumulative and by discrete age-intervals) | ≤360 days after birth
LRTI hospitalization (any cause) occurring ≤360 days after birth (first episode during the RSV season) (cumulative and by age-intervals) | ≤360 days after birth
ARI hospitalization (any cause) occurring ≤360 days after birth (first episode during the RSV season) (cumulative and by age-intervals) | ≤360 days after birth

OTHER OUTCOMES:
PCR-confirmed RSV-associated hospitalization stratified by: gestational age (GA) at delivery, GA at vaccination, time from vaccination to birth, with/without administration with other maternal vaccines, breastfeeding status & infant deprivation index | ≤360 days after birth
Infant & hospitalization characteristics (e.g. infant age at hospitalization, duration of stay in days, level of care, disease severity, death) among infants ≤360 days after birth with RSV-associated hospitalization & maternal ABYRSVO vaccination status | ≤360 days after birth
Relative risk of breakthrough RSV in infants born to mothers vaccinated with ABRYSVO by sex, gestational age at birth, low birth weight, deprivation index, ethnicity, time between vaccine and delivery, and maternal morbidity status. | ≤360 days after birth

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.